CLINICAL TRIAL: NCT00375557
Title: An Open Label, Randomized, Flexible Dose, 6-week Clinical Trial of the Safety and Efficacy of Divalproex ER vs Quetiapine in the Treatment of Behavioral Symptoms in the Elderly With Moderate to Severe Alzheimer's Dementia
Brief Title: Safety and Efficacy of Divalproex and Quetiapine in Elderly Alzheimer's Dementia Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Muhammad Aslamm, Associate Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 06-08-25-06
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Alzheimer's Disease; Dementia; Behavioral Symptoms
MeSH Terms: conditions — Alzheimer Disease; Dementia; Behavioral Symptoms | interventions — Valproic Acid; Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Quetiapine
  Interventions: Drug: Quetiapine
- 2 (Active Comparator): Divalproex ER
  Interventions: Drug: Divalproex ER

INTERVENTIONS:
Drug: Divalproex ER — Divalproex ER will be initiated on 250 mg/day, dosed once daily. The daily dose of Divalproex ER will be titrated up 250 mg each day based on patients' response and tolerability, not to exceed a maximum of 2000 mg/day.
  Other Names: Depakote ER
  Arms: 2
Drug: Quetiapine — Quetiapine will be initiated in 25 mg/day, with a variable dosing frequency (QD-TID). The daily dose of Quetiapine will be titrated up by 25-50 mg each day based on patients' response and tolerability, not to exceed a maximum of 750 mg/day.
  Other Names: Seroquel
  Arms: 1

SUMMARY:
The primary aim is to determine whether Divalproex ER or one of the atypical antipsychotics is more effective improving dementia related behavioral symptoms in patients with dementia, and evaluate the impact of such improvements on other clinical domains, such as quality of life, functional status.

DETAILED DESCRIPTION:
This clinical trial will be open label, flexible dose study of Divalproex ER vs Quetiapine for 6 weeks. Patients will be randomized to Divalproex ER vs Quetiapine outpatient / inpatient. The schedule of visits will include a screening, a baseline and 3 treatment visits / assessment. The End of Study/Early Termination visit will conclude the Trial. The safety follow-up visit will be scheduled only for the patients with unresolved Adverse Events detected prior or at the End of Study/Early Termination visit.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, men and women =/> 55 years of age.
2. Inpatient / Outpatients with diagnosis of Moderate to Severe probable Alzheimer's dementia as determined by the Structured Clinical Interview for DSM-IV.
3. Patients with a Mini Mental Status Examination scores between 3-15 at screening.
4. Patients and Care Giver/ Legal representative or Guardian who are able to comprehend and satisfactorily comply with protocol requirements.
5. Patient, Care Giver/ Legal representative or Guardian who signed the written informed consent given prior to entering any study procedure.
6. Patients who have been at least three month ongoing stable dose of cholinesterase enzyme inhibitors or memantine.

Exclusion Criteria:

1. Patients with a concurrent DSM-IV Axis I diagnosis in any of the following categories:

   1.1. Delirium, Amnestic and other Cognitive disorders 1.2. Lifetime Schizophrenia and other Psychotic Disorders 1.3. Lifetime Bipolar I Disorder 1.4. Bipolar 11 Disorder with an episode of hypomania within the last year 1.5. Alcohol or Substance Dependence or Abuse (excluding nicotine) in one month prior to the Screening Visit
2. Patients with a history of intolerance or hypersensitivity to Divalproex ER & Quetiapine.
3. Patients who have a history of seizures.
4. Patients who based on history or mental status examination have a significant risk of committing suicide.
5. Patients who are homicidal or violent and who are in the Investigator's opinion in significant imminent risk of hurting others.
6. Patients who have been treated with depot-neuroleptic within 3 months prior to the Baseline Visit.
7. Patients with a positive urine drug screen, unless proven to be prescribed for a short-term course of treatment. In these situations a urine drug screen must be repeated at least 7 days after the last dose of the prescription medication containing narcotics.
8. Patients who have participated in any clinical trial within one month prior to the Screening Visit, or in a clinical trial involving a psychotropic medication within the 3 months prior to the Screening Visit.
9. Patients who have a medical condition that, in the Investigator's opinion, would expose them to an increased risk of a significant adverse event or interfere with assessments of safety and efficacy during the course of the trial.
10. Patients with any current malignancy, or any clinically significant hematological, endocrine, cardiovascular, renal, hepatic, gastrointestinal or neurological disease (including any form of epilepsy). If there is a history of such disease but the condition has been stable for at least the past year and is judged by the investigator not to interfere with the patient's participation in the study, the patient may be included.
11. Patients with systolic blood pressure greater than 180 mm Hg or less than 90 mm Hg or diastolic blood pressure greater than 105 mm Hg or less than 50 mm Hg at the Screening visit.
12. Patients who test positive for Hepatitis B surface antigen or Hepatitis C antibody.
13. Patients whose laboratory values at the Screening visit will be 1.5 times greater than ULN.
14. Patients requiring concomitant treatment with any psychotropic drug (except zolpidem for sleep no more than 3x/week prn).
15. Patients who require concomitant therapy with any prohibited prescription.
16. Patients who are unable to speak, read, and understand English or are judged by the investigator to be unable or unlikely to follow the study protocol and complete all scheduled visits.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-10; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
The change from the Baseline to the End of the Study/Early Termination visit in the CMAI & Quality of life scale scores. | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Aslam, MD, Principal Investigator — University of Cincinnati/ VA Medical Center
Locations (1):
- Cincinnati VA Hospital, Cincinnati, Ohio, United States

REFERENCES:
- [Background] Profenno LA, Jakimovich L, Holt CJ, Porsteinsson A, Tariot PN. A randomized, double-blind, placebo-controlled pilot trial of safety and tolerability of two doses of divalproex sodium in outpatients with probable Alzheimer's disease. Curr Alzheimer Res. 2005 Dec;2(5):553-8. doi: 10.2174/156720505774932205. PMID 16375658